CLINICAL TRIAL: NCT05879627
Title: A Multicenter, Open Phase I Clinical Study to Evaluate the Safety, Tolerance and Pharmacokinetics of BAT8007 for Injection in Patients With Advanced Solid Tumors
Brief Title: To Evaluate the Safety, Tolerance and Pharmacokinetics of BAT8007 for Injection in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Collaborators: Zhejiang Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-8007-001-CR
Record Dates: First submitted 2023-02-07; First posted 2023-05-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 2 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 3 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 4 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 5 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 6 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 7 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection
- Cohort 8 (Experimental): BAT8007 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8007 for injection

INTERVENTIONS:
Drug: BAT8007 for injection — Intravenous infusion: once every three weeks.The infusion time in the first cycle is recommended to be ≥ 90 minutes. If no infusion reaction occurs, the subsequent cycle can be completed within 30~120 minutes.
  Other Names: Recombinant all human anti Nectin-4 monoclonal antibody for injection Exatecan conjugate

SUMMARY:
A multicenter, open phase I clinical study to evaluate the safety, tolerance and pharmacokinetics of BAT8007 for injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open, dose increasing and dose expanding Phase I clinical study. About 169~292 patients will be enrolled from research centers in China, the United States, Australia, etc. In the dose increasing stage, accelerated titration and "3+3" dose increasing design were used to explore the safety, tolerance and PK characteristics of BAT8007 for injection in patients with advanced solid tumors. During the dose increasing test, select the appropriate dose according to the previous study data for the extended study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (including the boundary value), regardless of gender;
* Sign the informed consent form voluntarily;
* Dose-climbing studies: cytologically or histologically confirmed patients with advanced solid tumors who failed standard therapy, had no standard therapy, were intolerant to standard therapy, or refused to receive standard therapy; Dose-expansion studies: Patients with cytologically or histologically confirmed locally advanced/metastatic urothelial carcinoma or other advanced or metastatic solid tumors with cytologically or histologically confirmed failure of standard therapy or intolerance to standard therapy (at least first-line systemic antitumor therapy).
* Patients in the dose increasing study must have an evaluable tumor focus, and patients in the dose expanding study must have at least one measurable tumor focus (according to RECIST 1.1 standard);
* The physical status score of the East American Cooperative Oncology Group (ECOG) is required to be 0 or 1;
* The investigator assessed that the expected survival period was ≥ 12 weeks;
* Prepare sufficient organ and bone marrow reserve function, and the definition is as follows: blood routine test (no blood component, cell growth factor support treatment and no drug to correct the number of blood cells within 14 days before the first administration), absolute neutrophil count (ANC) ≥ 1.5 × 109/L platelet count ≥ 90 × 109/L hemoglobin ≥ 90g/L coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (those not receiving anticoagulation therapy) can be included in patients receiving oral anticoagulation therapy with INR of 2-3; Subjects currently receiving intravenous or subcutaneous anticoagulation therapy must be excluded. Liver function: total bilirubin (TBIL) generally ≤ 1.5 × ULN； Hepatocellular carcinoma, liver metastasis ≤ 2 × ULN alanine aminotransferase (ALT), aspartate aminotransferase (AST) generally ≤ 2.5 × ULN； Hepatocellular carcinoma, liver metastasis ≤ 5 × ULN Renal function: serum creatinine ≤ 1.5 × ULN or serum creatinine clearance>60ml/min (Cockcroft Gault formula is adopted, see appendix)
* Female patients with fertility must have negative serum pregnancy test within 7 days before the first administration and be willing to take effective birth control/contraception methods to prevent pregnancy during the study period until 6 months after the last administration. Male patients must agree to take effective contraceptive methods during the study period until 6 months after the last administration of the drug; Postmenopausal women must be amenorrhoea for at least 12 months before they are considered infertile;
* We must agree to abide by the epidemic prevention regulations of the host country and region against COVID-19 novel coronavirus, and minimize the exposure to COVID-19 from the screening period to the end of the study (28 days of safety follow-up);
* Able to understand the test requirements, willing and able to follow the test and follow-up procedures.

Exclusion Criteria:

* Within 4 weeks before the first administration of the study drug, he received experimental drug treatment;
* Subjects who have received previous treatment with Nectin-4 or related target research drugs (not limited to antibody, ADC, etc.);
* Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first use of the study drug, except for the following: ① Nitrosourea or mitomycin C within 6 weeks before the first use of the study drug; ② Oral fluorouracil and small molecule targeted drugs were taken 2 weeks before the first use of the study drug or within 5 half lives of the drug (whichever is longer); ③ Within 2 weeks before the first use of the investigational drug, the systematic treatment of traditional Chinese medicine/Chinese patent medicine with clear anti-tumor effect and drugs with immunomodulatory effect (including but not limited to thymosin, interferon, interleukin, etc.); ④ Palliative radiotherapy was performed within 2 weeks before the first use of the study drug;
* After receiving any topoisomerase I inhibitor (such as irinotecan) in the past, there has been a drug related or unknown AE ≥ 3 levels (using CTCAE version 5.0 for grading);
* Before the first administration of the study drug, AE (CTCAE version 5.0) caused by previous anti-tumor treatment was still greater than grade 1, except for the following circumstances: a. alopecia; B pigmentation; c. The distal neurotoxicity caused by chemotherapy and radiotherapy can not be further recovered after judgment; d. Stable hypothyroidism after hormone replacement therapy;
* Patients who have undergone major surgery or have not recovered from surgery within 4 weeks before the first administration of the study drug, or have experienced significant trauma, or need to undergo elective surgery during the trial. Note: Those who have undergone minor surgery ≥ 28 days before screening must have fully recovered from the surgery before the first administration, except for the indwelling operation at the intravenous infusion port;
* Have a history of allograft cell or solid organ transplantation;
* Primary central nervous system tumor or symptomatic central nervous system metastasis (meningeal metastasis with or without symptoms must be excluded). Patients with asymptomatic or symptomatic central nervous system metastasis who have reached clinical control but are judged by the researcher to be stable can be included, but the following conditions must be met simultaneously: a The clinical symptoms were stable ≥ 4 weeks before the first administration; b. No evidence of progression of central nervous system disease was found in brain MRI enhancement within 4 weeks before the first administration; c. The antiepileptic drugs have been stopped at least 2 weeks before the first medication;
* In the dose expansion study, there were other active malignant tumors within 3 years before the first administration. Except for locally cured tumors (such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer or breast cancer in situ);
* The following cardiovascular diseases occurred within 6 months before the first drug use: symptomatic heart failure with NYHA grade of 2 or above, left ventricular ejection fraction (LVEF)<50%, unstable arrhythmia or unstable angina pectoris, myocardial infarction requiring treatment, pulmonary embolism Uncontrolled hypertension (this protocol is defined as systolic blood pressure > 160mmHg and/or diastolic blood pressure > 100mmHg after treatment, although the optimal antihypertensive treatment is used, and it is evaluated by the researcher as clinically significant). Note: 3 times of 12 lead ECG suggested that QTc interval extension>450 ms (male) or>470 ms (female) should be excluded; The patients with atrial fibrillation or paroxysmal supraventricular tachycardia that must be treated can be considered to be included after the investigator has assessed that the condition is stable;
* Suffering from any other disease, physical examination or laboratory examination results, which are not suitable for the use of the study drug according to the judgment of the investigator;
* Subjects who had previously suffered from non infectious pneumonia/pulmonary inflammation requiring glucocorticoid treatment, or currently suffered from interstitial lung disease (ILD), or failed to rule out ILD/pulmonary inflammation through imaging examination during the screening period;
* Untreated or under treatment tuberculosis subjects, including but not limited to tuberculosis; Those who have been treated with standardized anti tuberculosis treatment and confirmed to be cured by researchers can be included;
* Serious infection occurred within 4 weeks or active infection occurred within 2 weeks before the first medication;
* People infected with the following diseases: human immunodeficiency virus (HIV) infection; Active hepatitis B virus infected persons [hepatitis B surface antigen (HBsAg) is positive, and the detection of hepatitis B virus deoxyribonucleic acid (HBV-DNA) is>200 IU/ml or 103 copies/ml]; HCV infected persons [HCV antibody and viral ribonucleic acid (HCV RNA) detection results are positive]; Treponema pallidum antibody positive and RPR positive;
* Known hypersensitivity or delayed anaphylaxis to any component of the study drug;
* It is known that there has been ≥ grade 3 allergic reaction to macromolecular protein preparation/monoclonal antibody;
* Patients with uncontrollable pleural effusion, pericardial effusion or peritoneal effusion within 2 weeks before the first administration or who need drainage;
* Those with the following risk of thrombosis or bleeding:

  1. Cerebrovascular accident or transient ischemic attack occurred within 6 months before the first administration;
  2. There is a history of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months before the first administration (implanted venous infusion port or catheter derived thrombosis, or superficial venous thrombosis is not considered as "serious" thromboembolism);
  3. Any life threatening bleeding event or grade 3 or 4 gastrointestinal/variceal bleeding event requiring blood transfusion, endoscopy or surgery within 3 months before the first administration;
  4. Other diseases that the researchers believe have a high risk of bleeding or thrombosis in the future;
* Existence of any other serious underlying disease (such as Gilbert syndrome, unstably controlled diabetes, active gastric ulcer, unstably controlled convulsion, coagulation dysfunction with serious symptoms or signs);
* Known psychiatric diseases, drug abuse history, alcohol abuse history or drug abuse history, which affect the test results;
* Pregnant or lactating women or women or men preparing for childbirth;
* Those who have received any live attenuated vaccine within 4 weeks before the first administration of the study drug. About COVID-19 vaccination: the interval between COVID-19 vaccination and the first administration must be at least 14 days, and COVID-19 vaccination is not allowed during DLT observation. Some special cases can be included in the study with the consent of the medical supervisor;
* It is estimated that the patient's compliance to participate in this clinical study is insufficient or the investigator believes that there are other factors that are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | A minimum of 21 days after first dose of BAT8007
  number of subjects who experience DLT events during 21 days. Toxicity will be graded according to NCI CTCAE, Version 5.0.
Adverse Events (AEs) | AE needs continuous monitoring and evaluation from the first administration to 28 days after the last administration or before receiving new anti-tumor treatment.
  Incidence of treatment -related AEs as assessed by NCI CTCAE, Version 5.0.

SECONDARY OUTCOMES:
Anti-drug antibodies (ADA) | up to Cycle 3, each cycle is 14 days
  Level of ADA
neutralizing antibodies (NAb) | up to Cycle 3, each cycle is 14 days
  Level of NAb
Cmax | up to Cycle 3, each cycle is 14 days
  Level of Cmax
Tmax (Time to reach maximum serum concentration) | up to Cycle 3, each cycle is 14 days
  Level of Cmax
T1/2 (terminal half-life) | up to Cycle 3, each cycle is 14 days
  Level of T1/2
Systemic Clearance (CL) | up to Cycle 3, each cycle is 14 days
  Level of CL

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, PI, Principal Investigator — Medical Ethics Committee of Zhejiang Cancer Hospital
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No